CLINICAL TRIAL: NCT03621878
Title: Effect of Neural Mobilization Techniques on Pain, and Hip and Knee Range of Motion on Lumbosacral Radiculopathy Patients With Peripheral Sensitization
Brief Title: Effect of Neural Mobilization on Lumbosacral Radiculopathy Patients With Peripheral Sensitization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed Al-Ghamdi (Other)
Responsible Party: Sponsor-Investigator, Mohammed Al-Ghamdi, Physical Therapist, Imam Abdulrahman Bin Faisal University
Organization: Imam Abdulrahman Bin Faisal University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-2014-04-321
Record Dates: First submitted 2018-07-30; First posted 2018-08-09 (Actual); Results first posted 2019-07-22 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Radiculopathy
Keywords: Lumbosacral radiculopathy; peripheral sensitization; Neural mobilization; radicular LBP; slider; tensioner
MeSH Terms: conditions — Radiculopathy | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: both the examiner and the outcomes assessor where blinded to the participants groups. the primary investigator was also blind to the outcomes of each participant during the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Patients in this group had 6 sessions in 2 weeks of Transcutaneous Electric Nerve Stimulation (TENS).
  Interventions: Other: Transcutaneous Electrical Nerve Stimulation (TENS)
- Tensioner Group (Experimental): Patients in this group had 6 sessions in 2 weeks of TENS combined with neural mobilization exercises (Tensioner technique).
  Interventions: Other: Neural mobilization exercises -Tensioner technique
- Slider Group (Experimental): Patients in this group had 6 sessions in 2 weeks of TENS combined with neural mobilization exercises (Slider technique).
  Interventions: Other: Neural mobilization exercises -Slider technique

INTERVENTIONS:
Other: Neural mobilization exercises -Tensioner technique — Exercise aiming to lengthen the neural structure using more than one joint.
  Arms: Tensioner Group
Other: Neural mobilization exercises -Slider technique — Exercise aiming to slide/glide the neural structure using more than one joint.
  Arms: Slider Group
Other: Transcutaneous Electrical Nerve Stimulation (TENS) — Electrotherapy device aiming to decrease patient's symptoms.
  Other Names: Control
  Arms: Control group

SUMMARY:
The primary purpose of this study was to investigate the effects of slider and tensioner techniques on pain, hip and knee ROM in lumbosacral radiculopathy patients with peripheral sensitization. A secondary purpose was to evaluate the correlation between these outcomes measurements.

DETAILED DESCRIPTION:
Study design: Double-blind case-control trial. Methods: Fifty-one male lumbosacral radiculopathy patients with peripheral sensitization, were divided into one of the three groups: slider, tensioner, and control. The primary outcome measurements were visual analog scale (VAS) for pain, hip range of motion (ROM) during SLR test, and knee flexion ROM during slump test. The measurements were taken at baseline, after 1st, 3rd, and 6th session.

Statistical Analysis: A two-way mixed design analysis of variance (MANOVA) with post-hoc (Bonferonni Correction) was used to calculate the differences with Time (baseline, 1st,3rd,6th sessions) as a within-group factor and Group (control, slider, and tensioner) as a between-group factor. The effect size was calculated with Cohen's d. Pearson's correlation was used for correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lumbosacral radiculopathy with dominant peripheral sensitization
* patients with unilateral leg pain.
* patient S-LANSS score > 12,
* negative sensory and motor examination.
* positive neural tissue provocation tests (straight leg raising test, slump test).
* adult.
* pain duration of more than 3 months.

Exclusion Criteria:

* S-LANSS score ≥ 12,
* motor or sensory deficits,
* history of back or lower extremity surgeries,
* bilateral referred pain,
* patients with pacemakers, cardiovascular problems, epilepsy, active malignancy, dermatological conditions, and diminished pain sensation.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2018-03-30 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: patients in this group had 6 session of Transcutaneous Electric Nerve Stimulation in 2 weeks.
  Transcutaneous Electric Nerve Stimulation: electric current produced by a device to stimulate the nerves for pain management
- Tensioner Group: patients in this group had 6 session of TENS combined with Neural mobilization exercises -Tensioner technique in 2 weeks.
  Neural mobilization exercises -Tensioner technique: a maneuver was done to increase the tension by lengthening the neural structure
  Transcutaneous Electric Nerve Stimulation: electric current produced by a device to stimulate the nerves for pain management
- Slider Group: patients in this group had 6 session of TENS combined with Neural mobilization exercises -Slider technique in 2 weeks.
  Neural mobilization exercises -Slider technique: maneuver that produces a sliding motion between the neural tissues and the surrounding structures
  Transcutaneous Electric Nerve Stimulation: electric current produced by a device to stimulate the nerves for pain management
Period: Overall Study
Arm/Group | Control Group | Tensioner Group | Slider Group
Started (the data from subject whom completed the trials only was used in the statistical analysis and result) | 17 | 17 | 17
Completed | 17 | 17 | 17
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Tensioner Group | Slider Group | Total
Number analyzed (Participants) | 17 | 17 | 17 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.24 (9.49) | 33.53 (8.64) | 36.82 (8.01) | 36.86 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 17 | 17 | 17 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
body mass insex [Median (Standard Deviation); unit: Kg/m^2] | 27.08 (3.83) | 28.23 (6.04) | 28.19 (5.60) | 27.83 (5.16)
Pain [Mean (Standard Deviation); unit: Centimeters] — visual analog scale was used to measure pain intensity in the baseline measurement. this scale is a 10 cm line where patients chose from 0 to 10 (when 0 mean no pain and 10 mean maximum pain)
  Centimeters | 5.63 (1.75) | 5.09 (1.95) | 5.05 (2.15) | 5.26 (1.93)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale
Description: Visual analog scale was used to measure pain intensity. This scale is a 10 cm line where patients chose from 0 to 10 (when 0 mean no pain and 10 mean maximum pain)
Time Frame: The measurements were taken at days "0,1,5,12"
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Control Group | Slider Group | Tensioner Group
Number analyzed (Participants) | 17 | 17 | 17
Centimeters
  Basline | 5.638 (1.75762) | 5.050 (2.15029) | 5.094 (1.95015)
  After 1st Day | 4.894 (1.86001) | 4.759 (1.99125) | 3.576 (2.22810)
  After 5th Day | 5.100 (1.87508) | 3.556 (2.21613) | 2.606 (2.02005)
  After 12th Day | 4.665 (1.74676) | 2.626 (2.23538) | 2.082 (1.56734)

2. Primary Outcome: Hip Flexion Range of Motion (Symptomatic Side)
Description: Change in Hip flexion range of motion during straight leg raising (symptomatic side)
Time Frame: The measurements were taken at days "0,1,5,12"
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Control Group | Slider Group | Tensioner Group
Number analyzed (Participants) | 17 | 17 | 17
degrees
  Baseline | 51.82 (15.314) | 57.71 (16.042) | 46.29 (16.243)
  After 1st Day | 58.53 (13.884) | 63.59 (15.452) | 58.88 (16.714)
  After 5th Day | 59.24 (14.338) | 67.47 (15.412) | 62.82 (13.956)
  After 12th Day | 57.71 (17.944) | 74.41 (22.327) | 68.59 (12.555)

3. Primary Outcome: Knee Flexion Range of Motion (Symptomatic Side)
Description: Change in Knee flexion range of motion during slump (symptomatic side)
Time Frame: The measurements were taken at days "0,1,5,12"
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Control Group | Slider Group | Tensioner Group
Number analyzed (Participants) | 17 | 17 | 17
degrees
  Baseline | 52.29 (17.395) | 45.647 (18.435) | 47.059 (14.545)
  After 1st Day | 49.41 (17.603) | 31.294 (12.133) | 34.824 (15.509)
  After 5th Day | 48 (14.018) | 31.412 (14.590) | 31.765 (14.342)
  After 12th Day | 47 (16.733) | 26.882 (15.419) | 64.47 (25.529)

4. Primary Outcome: Hip Flexion Range of Motion (Asymptomatic Side)
Description: Change in Hip Flexion Range of Motion During Straight Leg Raising (Asymptomatic Side)
Time Frame: The measurements were taken at days "0,1,5,12"
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Control Group | Slider Group | Tensioner Group
Number analyzed (Participants) | 17 | 17 | 17
degrees
  Baseline | 70.00 (15.313) | 71.824 (20.467) | 63.59 (15.407)
  After 1st Day | 69.41 (17.044) | 70.82 (20.944) | 69.12 (13.114)
  After 5th Day | 71.12 (11.146) | 74.12 (18.721) | 72.12 (11.033)
  After 12th Day | 73.06 (12.920) | 74.88 (19.251) | 72.47 (10.869)

5. Primary Outcome: Knee Flexion Range of Motion (Asymptomatic Side)
Description: Change in Knee flexion range of motion during slump (Asymptomatic side)
Time Frame: The measurements were taken at days "0,1,5,12"
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Control Group | Slider Group | Tensioner Group
Number analyzed (Participants) | 17 | 17 | 17
degrees
  Baseline | 31.1176 (19.70052) | 31.7059 (12.01439) | 28.8824 (18.01001)
  After 1st Day | 30.41 (22.319) | 24.06 (13.831) | 26.06 (14.528)
  After 5th Day | 28.94 (18.216) | 28.76 (19.250) | 23.88 (13.453)
  After 12th Day | 24.88 (17.517) | 22.29 (16.669) | 20.35 (12.639)

ADVERSE EVENTS:
Time Frame: data was collected in around 3 years
Description: no participants was in risk of mortality or Serious Adverse Events because the participants in this study ware patients with mild low back pain and and all the treatment we used ware gentle and without any serious adverse effects.
Arm/Group | Control Group | Tensioner Group | Slider Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT03621878/Prot_SAP_000.pdf